CLINICAL TRIAL: NCT02538926
Title: A Phase II Study of Dose-Adjusted Etoposide, Prednisone, Vincristine, Cyclophosphamide, and Doxorubicin Plus Asparaginase (DA-EPOCH-A) for Adults With Acute Lymphoblastic Leukemia/Lymphoma
Brief Title: Etoposide, Prednisone, Vincristine Sulfate, Cyclophosphamide, and Doxorubicin Hydrochloride With Asparaginase in Treating Patients With Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drugs unavailable
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9459; NCI-2015-01402 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CC9459; 9459 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: B Acute Lymphoblastic Leukemia; B Lymphoblastic Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent B Lymphoblastic Lymphoma; Recurrent T Lymphoblastic Leukemia/Lymphoma; Refractory B Lymphoblastic Lymphoma; Refractory T Lymphoblastic Lymphoma; T Acute Lymphoblastic Leukemia; T Lymphoblastic Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Leyk; Cyclophosphamide; Doxorubicin; Etoposide; Imatinib Mesylate; Prednisone; deltacortene; prednylidene; Rituximab; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (DA-EPOCH-A) (Experimental): Patients receive etoposide, doxorubicin hydrochloride, and vincristine sulfate IV continuously over days 1-4, cyclophosphamide IV over 1 hour on day 5, and prednisone PO BID on days 1-5. Patients also receive asparaginase IM or IV over 1-2 hours every 2-3 days, beginning day 7 of each course. Patients who are CD20 positive and Philadelphia chromosome negative also receive rituximab IV on day 1 or 5. Patients who are Philadelphia chromosome positive also receive imatinib mesylate PO on days 1-14. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Asparaginase; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Imatinib Mesylate; Other: Laboratory Biomarker Analysis; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Asparaginase — Given IM or IV
  Other Names: ASP-1; Asparaginase II; Asparaginase-E.Coli; Colaspase; Elspar; Kidrolase; L-Asnase; L-ASP; L-Asparaginase; L-Asparagine Amidohydrolase; Laspar; Lcf-ASP; Leucogen; Leunase; MK-965; Paronal; Re-82-TAD-15; Serasa
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Imatinib Mesylate — Given PO
  Other Names: CGP 57148; CGP57148B; Gleevec; Glivec; STI 571; STI-571; STI571
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar BI 695500; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; RTXM83
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well etoposide, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride with asparaginase work in treating patients with acute lymphoblastic leukemia or lymphoblastic lymphoma. Drugs used in chemotherapy, such as etoposide, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Asparaginase breaks down the amino acid asparagine and may block the growth of tumor cells that need asparagine to grow. Giving combination chemotherapy with asparaginase may work better in treating patients with acute lymphoblastic leukemia or lymphoblastic lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of dose-adjusted etoposide, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride plus asparaginase (DA-EPOCH-A) in adults with acute lymphoblastic leukemia/lymphoma (ALL).

SECONDARY OBJECTIVES:

I. To evaluate the safety and feasibility of this regimen.

OUTLINE:

Patients receive etoposide, doxorubicin hydrochloride, and vincristine sulfate intravenously (IV) continuously over days 1-4, cyclophosphamide IV over 1 hour on day 5, and prednisone orally (PO) twice daily (BID) on days 1-5. Patients also receive asparaginase intramuscularly (IM) or IV over 1-2 hours every 2-3 days, beginning day 7 of each course. Patients who are cluster of differentiation (CD)20 positive and Philadelphia chromosome negative also receive rituximab IV on day 1 or 5. Patients who are Philadelphia chromosome positive also receive imatinib mesylate PO on days 1-14. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of either B- or T-cell acute lymphoblastic leukemia or lymphoblastic lymphoma that is either:

  * Arm A: Initially diagnosed at age 40 or later, OR
  * Arm B: Relapsed after or failed to respond to >= 1 previous chemotherapy regimen
* The regimen under study must constitute a reasonable therapeutic option
* Presence of >= 5% abnormal blasts in the bone marrow
* Patients with prior allogeneic hematopoietic cell transplantation (HCT) must be at least 90 days post-HCT and must be on =< 20 mg of prednisone (or equivalent dose of an alternative corticosteroid) for treatment/prevention of graft-vs-host disease
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN; unless attributable to Gilbert's disease or other causes of inherited indirect hyperbilirubinemia, at which point total bilirubin must be =< 2.5 x ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN
* Note: Patients with liver test abnormalities attributable to hepatic involvement by ALL will be permitted if the total bilirubin is =< 3.0 x ULN and ALT/AST are =< 5.0 x ULN
* Creatinine =< 1.5 mg/dL; however, patients with a creatinine > 1.5 mg/dL but with a calculated creatinine clearance of > 60 ml/min, as measured by the Modification of Diet in Renal Disease (MDRD) equation, will be eligible
* Measurement of left ventricular ejection fraction (LVEF) should be performed in patients with prior anthracycline exposure or known history of arrhythmia or structural heart disease; in these cases, LVEF must be >= 40%
* As patients with ALL frequently have cytopenias, no hematologic parameters will be required for enrollment or to receive the first cycle of treatment; however, adequate recovery of blood counts will be required to receive subsequent cycles
* Per good clinical practice, any toxicity related to prior therapies that, in the opinion of the investigator, would potentially be worsened with DA-EPOCH-A +/- imatinib (imatinib mesylate) +/- rituximab, should be resolved to grade 1 or less
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Women of childbearing potential must have a negative pregnancy test and must agree to the use of effective contraception while on treatment; men must also agree to the use of effective contraception while on treatment
* Ability to give informed consent and comply with the protocol
* Anticipated survival of at least 3 months

Exclusion Criteria:

* Patients with Burkitt lymphoma/leukemia
* Patients must not have received chemotherapy within 14 days of enrollment, with the two following exceptions:

  * Routine systemic maintenance therapy (e.g., Abelson murine leukemia viral oncogene homolog 1 [ABL] kinase inhibitor, methotrexate, 6-mercaptopurine, vincristine, etc.) and intrathecal/intraventricular therapy
  * Systemic therapy for the acute management of hyperleukocytosis or acute symptoms (e.g., corticosteroids, cytarabine, etc.)
* May not have prior malignancies unless the expected survival is at least 2 years
* For patients with Philadelphia chromosome positive (Ph+) ALL, they must not have progressed within 3 months of receiving imatinib or have a documented ABL kinase mutation known to confer resistance to imatinib (e.g., T315I)
* Patients with persistent grade 2 or higher peripheral sensory or motor neuropathy of any cause
* Patients with isolated extramedullary disease or with parenchymal central nervous system (CNS) disease
* Known hypersensitivity or intolerance to any of the agents under investigation
* Human immunodeficiency virus (HIV) positive or evidence of infection with hepatitis B or C virus, as defined by any of the following criteria (if patients have not previously been tested for the following, these will be conducted during screening):

  * HIV antibody positive
  * Hepatitis B surface antigen or core antibody positive
  * Hepatitis C antibody positive
* Other medical or psychiatric conditions that in the opinion of the investigator would preclude safe participation in the protocol
* May not be pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Complete minimal residual disease response rate | Up to 5 years
  A Simon two-stage optimum design will be used to define success of this treatment in the two subgroups of patients.
Overall response rate (complete response + partial response) | Up to 5 years
  A Simon two-stage optimum design will be used to define success of this treatment in the two subgroups of patients.
Overall survival | From time of initiation of study therapy to up to 5 years
  A Simon two-stage optimum design will be used to define success of this treatment in the two subgroups of patients.
Progression-free survival | From time of initiation of study therapy to up to 5 years
  A Simon two-stage optimum design will be used to define success of this treatment in the two subgroups of patients.

SECONDARY OUTCOMES:
Incidence of adverse events, graded using the National Cancer Institute Common Terminology Criteria for Adverse Events | Up to 30 days post-treatment, or until patient receives an alternative anti-cancer therapy, whichever date comes first

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Cassaday, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States